CLINICAL TRIAL: NCT04690543
Title: Comparison of Length Gain Between Square Flap and Z-plasty in Post Burn Contracture Release
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Aiman Naseem, FCPS trainee, plastic surgery, DUHS, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANaseem
Record Dates: First submitted 2020-12-25; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Burn Scar

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- z-plasty (Active Comparator): Z-plasty: It will be defined as a local transposition flap that will be used to improve the functional and cosmetic appearance of scars. It will be involved creating two triangular flaps of equal dimensions that will be transposed.
  Interventions: Procedure: z-plasty
- square flap (Experimental): Square flap: It will be defined as is another local transposition flap which will be used for release of contractures. Square will be marked on one side of the contracture, and two triangles will be marked on the other side, with the length of all the flaps equal, which will be then transposed.
  Interventions: Procedure: square flap

INTERVENTIONS:
Procedure: z-plasty — Z-plasty: It will be defined as a local transposition flap that will be used to improve the functional and cosmetic appearance of scars. It will be involved creating two triangular flaps of equal dimensions that will be transposed.
  Arms: z-plasty
Procedure: square flap — Square flap: It will be defined as is another local transposition flap which will be used for release of contractures. Square will be marked on one side of the contracture, and two triangles will be marked on the other side, with the length of all the flaps equal, which will be then transposed.
  Arms: square flap

SUMMARY:
the purpose of this study is to compare the gain in length after postburn contracture release using two different techniques, the more commonly practised z - plasty and relatively newer technique, square flap

ELIGIBILITY:
Inclusion Criteria:- • Both genders.

* Joints supple.
* Linear contracture bands.
* Age between 5years to 50 years.
* Surrounding non scarred skin.
* Contractures of axilla, cubital fossa, popliteal fossa and digits.

Exclusion Criteria:

* Deep burns.

  * Joint contractures.
  * Surrounding skin scarred.
  * Broad, irregular contracture.
  * Neck, Perineal, wrist or toe contractures

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
gain in length | 3 weeks
  calculation of the gain in length achieved after the release of post burn contrature

CONTACTS AND LOCATIONS:
Overall Officials: Aiman Naseem, Principal Investigator — DUHS

IPD SHARING:
Plan to Share IPD: No